CLINICAL TRIAL: NCT00963196
Title: Supplementation of Antidepressants With Fatty Acid Therapy
Brief Title: Study of Supplementation of Antidepressants With Fish Oil to Improve Time to Clinical Response
Acronym: SADFAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: End of allotted time for subject recruiting.
Sponsor: University of Virginia (Other)
Responsible Party: Anita Clayton MD, University of Virginia Department of Psychiatry and Neurobehavioral Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14503
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- One unsuccessful trial (Active Comparator): Patients with one unsuccessful previous antidepressant trial
  Interventions: Dietary Supplement: Omega-3 fatty acid; Drug: Bovine gelatin capsules
- One successful trial (Active Comparator): Patients with one previous successful antidepressant trial
  Interventions: Dietary Supplement: Omega-3 fatty acid; Drug: Bovine gelatin capsules
- No previous trial (Active Comparator): Patients with no prior antidepressant therapy
  Interventions: Dietary Supplement: Omega-3 fatty acid; Drug: Bovine gelatin capsules

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — 2400mg daily of fish oil containing 1440mg combined EPA and DHA for 12 weeks
Drug: Bovine gelatin capsules — Bovine gelatin capsules that appear similar to active drug acting as placebo.

SUMMARY:
This study will be a randomized controlled trial set in an outpatient clinic, involving patients with major depressive disorder, who will be treated with antidepressant therapy, which will be individually agreed upon by the subject and his or her physician. Patients will be randomized to receive either placebo or fish oil capsules containing eicosapentaenoic acid (EHA) and docosahexaenoic acid (DHA) in addition to their antidepressant medication. Subjects will complete a brief dietary and exercise habits survey at the beginning of the trial to take into account lifestyle factors that may be significant in symptom resolution. Their progress will be monitored over a period of twelve weeks, with standardized rating scales completed by subjects and treating physicians. At the end of the study, scores will be compared between groups to look for differences in timing and degree of symptom improvement to analyze whether improvement occurred faster in the group receiving essential fatty acids (EFAs) than in the one receiving placebo. The primary hypothesis is that supplementation of antidepressant therapy with omega-3 fatty acids will decrease the lag period between the start of therapy and the time of clinically significant symptom improvement. A secondary hypothesis is that the results of this study will be consistent with numerous previous studies showing improvement in symptom control in major depressive disorder when antidepressants are supplemented with omega-3 fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder.
* Allowed comorbidities: Dysthymia, Anxiety Disorders.
* 18 years old or older.
* Males + Females.
* English-speaking.
* Women of reproductive age must be on adequate birth control, either oral contraceptives or using condoms or other barrier methods with spermicidal agents.
* Subjects may be undergoing psychotherapy, but must maintain current psychotherapy status. Must not start therapy if not already in therapy. If in therapy, must have received at least 6 sessions prior to entering the study.
* Subjects may continue taking herbals or supplements during the study, but they may not start any new herbals or supplements during the study.

Exclusion Criteria:

* 2 or more failed trials of antidepressants (adequate dose and duration, and documented).
* Substance dependence in the past 6 months.
* Current substance use or abuse (MJ, benzodiazepines, narcotics). If BZD use, patient must be tapered off and wait 1 month before being included in the trial.
* Psychosis.
* Bipolar Affective Disorder Type I, II or NOS.
* Pregnancy (current or planned).
* Unstable medical illness (pt has to be stable for at least 3 months, and may be excluded per investigator discretion).
* Dementia.
* Mental retardation.
* Traumatic Brain Injury.
* History of Stroke.
* History of seizure disorder.
* Electroconvulsive therapy within past 6 months.
* If, at the investigator's discretion, it is suspected that the subject will likely not comply with the study protocol.
* Imminent risk for suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in MADRS and PHQ-9 scores occurs in a shorter period of time in the intervention group versus the placebo group. | 12 weeks

SECONDARY OUTCOMES:
Subjects in the intervention group experience greater reduction of scores in MADRS and PHQ-9 than the placebo group. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anita H Clayton, MD, Principal Investigator — University of Virginia
Locations (1):
- UVA Psychiatry Outpatient Clinic, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Hallahan B, Garland MR. Essential fatty acids and mental health. Br J Psychiatry. 2005 Apr;186:275-7. doi: 10.1192/bjp.186.4.275. No abstract available. PMID 15802681
- [Background] Hallahan B, Garland MR. Essential fatty acids and their role in the treatment of impulsivity disorders. Prostaglandins Leukot Essent Fatty Acids. 2004 Oct;71(4):211-6. doi: 10.1016/j.plefa.2004.03.006. PMID 15301790
- [Background] Hibbeln JR. Fish consumption and major depression. Lancet. 1998 Apr 18;351(9110):1213. doi: 10.1016/S0140-6736(05)79168-6. No abstract available. PMID 9643729
- [Background] Gesch CB, Hammond SM, Hampson SE, Eves A, Crowder MJ. Influence of supplementary vitamins, minerals and essential fatty acids on the antisocial behaviour of young adult prisoners. Randomised, placebo-controlled trial. Br J Psychiatry. 2002 Jul;181:22-8. doi: 10.1192/bjp.181.1.22. PMID 12091259
- [Background] Pischon T, Hankinson SE, Hotamisligil GS, Rifai N, Willett WC, Rimm EB. Habitual dietary intake of n-3 and n-6 fatty acids in relation to inflammatory markers among US men and women. Circulation. 2003 Jul 15;108(2):155-60. doi: 10.1161/01.CIR.0000079224.46084.C2. Epub 2003 Jun 23. PMID 12821543
- [Background] Stoll AL, Severus WE, Freeman MP, Rueter S, Zboyan HA, Diamond E, Cress KK, Marangell LB. Omega 3 fatty acids in bipolar disorder: a preliminary double-blind, placebo-controlled trial. Arch Gen Psychiatry. 1999 May;56(5):407-12. doi: 10.1001/archpsyc.56.5.407. PMID 10232294
- [Background] Tanskanen A, Hibbeln JR, Hintikka J, Haatainen K, Honkalampi K, Viinamaki H. Fish consumption, depression, and suicidality in a general population. Arch Gen Psychiatry. 2001 May;58(5):512-3. doi: 10.1001/archpsyc.58.5.512. No abstract available. PMID 11343534
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851